CLINICAL TRIAL: NCT01132872
Title: PET Whole Body Distribution Studies Using the 5-HT1A Agonist, [11C]CUMI
Brief Title: PET Whole Body Distribution Studies Using [11C]CUMI
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100110; 10-M-0110
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-04-12

CONDITIONS: Depression; Major Depression; Unipolar Depression; Anxiety Disorder; Anxiety Disorders
Keywords: Serotonin 1A Receptor; Positron Emission Tomograhy (PET); Dosimetry; Healthy Volunteer; HV
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Depressive Disorder; Anxiety Disorders

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Researchers studying new treatments for major depressive disorder are looking at how medications to treat depression act on the brain chemical serotonin, which interacts with specific serotonin receptors on brain cells. New methods of studying serotonin receptors in the brain may help provide a better understanding of depression and treatment options.
* A new radioactive chemical called [11C]CUMI may be useful for studying serotonin receptors in the brain. By using positron emission tomography (PET) scanning to see how [11C]CUMI bonds with serotonin receptors, researchers will investigate whether [11C]CUMI can be used to study depression and how antidepressant medications work.

Objectives:

- To determine the usefulness of [11C]CUMI as a method of studying serotonin receptors in the brain.

Eligibility:

- Healthy individuals between 18 and 65 who have no history of psychiatric illness.

Design:

* This study requires 8 outpatient visits to the NIH clinic.
* Visit 1: Participants will have a full physical examination and medical history, as well as a psychiatric evaluation and questions about alcohol and drug use. Other tests will include blood and urine samples and an electrocardiogram (EKG). Testing will take approximately 3 hours.
* Visit 2: Participants will have a magnetic resonance imaging (MRI) scan to evaluate brain function and activity.
* Visit 3: Participants will have a PET scan, in which a small amount of the radioactive chemical [11C]CUMI will be injected through an intravenous (IV) catheter, and will have another IV line put in place to draw regular blood samples during the scan. The scan will last approximately 4 hours.
* Visits 4-8: Participants will have regular blood tests after the scan between days 1-3 and at about weeks 1, 2, 3, and 4. The blood tests will check muscle, heart, and liver function.

DETAILED DESCRIPTION:
Eighteen million people in the United States are currently suffering from Major Depressive Disorder, which is characterized by episodes of low mood, poor self attitude and poor vitality. Of those suffering from Major Depressive Disorder (MDD), only one third completely improve, but even among these cases, there is a waiting period of several weeks or more during which antidepressants take effect. Our inability to adequately treat MDD is evident in its being ranked number one in Disability Adjusted Life Years (DALY) among persons aged 15-44. Given this profound burden, improving our understanding of the molecular basis of MDD is of utmost importance in the development of novel antidepressant medications.

Serotoninergic neurotransmission is implicated in MDD, as demonstrated by the relative success of selective serotonin reuptake inhibitors (SSRIs). SSRIs block the reuptake of serotonin through the serotonin transporter, which then increases serotonin at the synaptic cleft. Serotonin then binds to 5-HT(1A) receptors, which are G-protein coupled receptors that are present both presynaptically and postsynaptically. Presynaptically, these receptors act as autoinhibitory receptors, triggering decreased firing rates and decreased serotonin release. This autoinhibitory mechanism is believed to be the reason why patients experience a delay in symptomatic improvement after initiation of SSRIs. Serotonin binding to postsynaptic receptors mediates symptomatic improvement of depression. Multiple positron emission tomography (PET) studies on 5-HT(1A) have been published. However, none of these studies use 5-HT(1A) agonists, which are specific for the high affinity, G-protein coupled and active state of the 5-HT(1A) receptor. We would therefore like to establish the use of the 5-HT(1A) radiolabelled agonist, [(11)C]CUMI, here at NIH.

The purpose of this study is to perform whole body PET studies in healthy volunteers in order to estimate radiation absorbed doses for [(11)C]CUMI. Future experiments will include studies on Major Depressive Disorder.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Subjects must be adults between 18-65 years old.
  2. Subjects must be able and willing to give written informed consent.

EXCLUSION CRITERIA:

1. With the exception of substance abuse disorders, any past or current Axis I diagnosis as assessed by clinical interview which may include the SCID-NP. With regard to substance abuse, we will allow a history of substance abuse so long as criteria for substance dependence are not met, and the episode(s) of substance abuse occurred over 1 year prior to study enrollment.
2. Any prior use of Lysergic acid diethylamide (LSD).
3. Use of ecstasy more than 3 times in a lifetime.
4. Any history of psychotic symptoms.
5. If female, any history of Premenstrual Dysphoric Disorder (PMDD), because PMDD has been shown to correlate with changes in 5-HT1A distribution in brain.
6. In women, irregular menses such that the subject will not know the phase of the menstrual cycle at time of scanning.
7. Clinically significant laboratory abnormalities.
8. Psychotropic medication use (including benzodiazepines and illicit drugs) during the 28 days (42 day for fluoxetine) prior to the PET scan.
9. Serious medical problems including but not limited to chronic neurological disease such as multiple sclerosis, autoimmune diseases or any cardiopulmonary disease that would increase risks associated with sedation.
10. Positive HIV status.
11. Head trauma resulting in a period of unconsciousness lasting longer than 10 minutes.
12. History of fetal alcohol syndrome or other neurodevelopmental disorder.
13. Recent exposure to radiation (i.e., PET from other research) which when combined with this study would be above the allowable limits.
14. Positive urine drug screen.
15. Inability to lie flat on camera bed for about 2.5 hours.
16. Pregnancy at time of scan (beta HCG will be measured in all female patients within 24 hours of scan and must be negative).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-04-30; Study Completion 2012-04-12

CONTACTS AND LOCATIONS:
Overall Officials: Marta Gozzi, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Alpert JE, Franznick DA, Hollander SB, Fava M. Gepirone extended-release treatment of anxious depression: evidence from a retrospective subgroup analysis in patients with major depressive disorder. J Clin Psychiatry. 2004 Aug;65(8):1069-75. PMID 15323591
- [Background] Amsterdam JD. Gepirone, a selective serotonin (5HT1A) partial agonist in the treatment of major depression. Prog Neuropsychopharmacol Biol Psychiatry. 1992 May;16(3):271-80. doi: 10.1016/0278-5846(92)90079-t. PMID 1350353
- [Background] Amsterdam JD, Brunswick DJ, Gibertini M. Sustained efficacy of gepirone-IR in major depressive disorder: a double-blind placebo substitution trial. J Psychiatr Res. 2004 May-Jun;38(3):259-65. doi: 10.1016/j.jpsychires.2003.10.005. PMID 15003431